CLINICAL TRIAL: NCT00525096
Title: A Multicenter Randomized Phase III, Double-blind Study Comparing Efficacy of the Association of Exemestane and Celecoxib Versus Exemestane and Placebo in Menopausal Patients With Metastatic Breast Cancer.
Brief Title: Exemestane + Celecoxib vs Exemestane + Placebo in Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Benedicte VOTAN, ARCAGY-GINECO
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CELAROM
Record Dates: First submitted 2007-09-03; First posted 2007-09-05 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Celecoxib; exemestane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Aromasin + placebo in place of Celebrex
  Interventions: Drug: placebo; Drug: Exemestane
- Celebrex (Experimental): Aromasin + Celebrex
  Interventions: Drug: Celecoxib; Drug: Exemestane

INTERVENTIONS:
Drug: placebo — 2 tablets twice a day per os
  Arms: Placebo
Drug: Celecoxib — 2*200 mg tablets twice a day per os
  Other Names: Celebrex
  Arms: Celebrex
Drug: Exemestane — Exemestane 25 mg per day per os
  Other Names: Aromasin

SUMMARY:
To discover if the adding of a coxib increases the efficacy of the Aromasine.

ELIGIBILITY:
Inclusion Criteria:

* Femal patient aged > 18 years
* Histologically proven breast cancer
* Menopausal patient according to the following definition:

  * amenorrhoea > 1 year or menopause affirmed by a rate of oestradiol or hypophyseal gonadotrophin
  * surgical ovariectomy
  * treatment by LHRH analog
  * ovarian suppression by radiotherapy
  * amenorrhoea induced by chemotherapy > 1 year
* Oestradiol and/or progesterone positive receptors
* Presence of one or several metastatic lesion:

  * mesurable lesion
  * bone metastase were detected by bone scintigraphy
* Patient who can have received:

  * Adjuvant chemotherapy and/or hormonotherapy (Tamoxifen)
  * Metastatic Treatment by chemotherapy
* PS < 2
* Adequate biological values
* Patient who has clearly given her consent by signing on informed consent form prior to participation

Exclusion Criteria:

* Patient previously treated with hormonotherapy in metastatic phase
* Antecedent of treatment with aromatase inhibitors
* local relapse (with the exception of cutaneous thoracic nodes)
* Patient with only one metastatic lesion like: pleurisy , ascites, lung Lymphangitis carcinomatosa

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2003-07; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 5 years

SECONDARY OUTCOMES:
Objective response rate | 6 months
Quality Of Life + pain | 6 months
Overall survival | 5 years
Tolerance | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gilles FREYER, PhD, Principal Investigator — Centre Hospitalier Lyon Sud - France